CLINICAL TRIAL: NCT05853276
Title: Effectiveness of Brush DJ App to Improve Oral Hygiene Compliance in Patients With Fixed Orthodontic Appliances - Randomised Controlled Study.
Brief Title: Effectiveness of Brush DJ App in Improving Oral Hygiene Compliance of Fixed Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IMU University, Malaysia (Other)
Responsible Party: Principal Investigator, Shilpa Gunjal, Dr, IMU University, Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IMU
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Gingivitis
Keywords: Gingival index; Plaque index; Fixed orthodontic appliance; Mobile application; Oral hygiene
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This group downloads and uses Brush DJ app. Reminders are sent through this app to brush their teeth and along with this oral hygiene instructions are also given.
  Interventions: Behavioral: Brush DJ app
- Control group (No Intervention): This group receives standard oral hygiene instructions

INTERVENTIONS:
Behavioral: Brush DJ app — Brush DJ app is a mobile app which can be freely downloaded. This app was chosen as part of the intervention as it was recognized by the NHS to reduce the risk of gum disease and tooth decay among its users. This app was built around the info given in the public health England Delivering Better Oral Health Toolkit.
  Arms: Intervention group

SUMMARY:
In this day and age, smartphones are occupying big portions of our lives. Expanding development of mobile applications focusing on delivering behavioral health intervention have intrigued us to know better about their efficacy.

Hence the present study was conducted to determine the effectiveness of the Brush DJ app on improving the oral hygiene compliance of patients wearing fixed orthodontic appliances by assessing their gingival status.

Null hypothesis: There was no difference in the gingival status and oral hygiene status of patients between verbal oral hygiene instructions and oral hygiene instructions using the Brush DJ app.

Research hypothesis: There was a difference in the gingival status and oral hygiene status of patients between verbal oral hygiene instructions and oral hygiene instructions using the Brush DJ app

DETAILED DESCRIPTION:
The participants are randomly distributed into two groups where Group I receive only standard oral hygiene instruction and Group II receive reminders via Brush DJ mobile application in addition to standard oral hygiene instructions. For the standard oral hygiene protocol received by participants of both groups, all of them are instructed to use soft-bristled toothbrushes, fluoridated toothpaste and interdental toothbrush or super floss. Proper oral hygiene education is provided to all the participants with the following 2-minute-long combined brushing technique.

For the evaluation of oral hygiene compliance of each orthodontic patient in each group, the gingival index according to Loë and Silness and Silness and Loe plaque index are measured at baseline (T0), 4th week (T1) and 8th week (T2). These indices are one of the standardized indicators of gingival health as it provides quantitative evaluation of the gingival status. GI and PI scores are measured by a single investigator who is calibrated. The reliability assessed by the intraclass correlation coefficient (ICC) suggested good agreement (0.85 & 0.88) for GI and PI respectively.

Data will be collected, cleaned, coded before doing the statistical analysis. The data will be checked for the range of Mean gingival index and Plaque index which should be within the range.

Sample size: The sample size was calculated to be 30 in each group, assuming a power of 80%, confidence interval of 95%, standard deviation (SD) of 0.5 and the aim of finding a 0.3 difference in the groups' means. All 60 volunteers were assessed for their eligibility before their participation.

ELIGIBILITY:
Inclusion Criteria:

1. participants who have smartphones with Android version ≥ 4.0.3 or IOS version ≥ 9 operating systems
2. participants willing to comply with given oral hygiene instructions
3. participants without periodontal disease and /or dental caries at the study onset
4. participants who receive their orthodontic appliances within one year after onset of study.

Exclusion Criteria:

1. participants with any mental and physical disability or craniofacial disorders
2. participants with enamel or dentin dysplasia
3. participants taking medications which affects plaque accumulation such as antibiotics or antibacterial mouth rinses
4. Participants with periodontal disease or dental caries at the onset of study.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Plaque index by Sillness and Loe | 12 weeks
  Reduction in the mean plaque index scores
Gingival index by Loe and Silness | 12 weeks
  Reduction in the mean gingival index scores

CONTACTS AND LOCATIONS:
Overall Officials: Shilpa Gunjal, PhD, Principal Investigator — IMU
Locations (1):
- IRDI, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No